CLINICAL TRIAL: NCT06042491
Title: The STRIVE Before Surgery Pilot Trial: a Vanguard Pragmatic Multicenter Randomized Trial of Structured TRaining to Improve Fitness in a Virtual Environment (STRIVE) Before Surgery
Brief Title: The STRIVE Before Surgery Pilot Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTO - 4479
Record Dates: First submitted 2023-08-10; First posted 2023-09-18 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Surgery-Complications; Disability Physical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Group allocation will not be indicated in data analyzed by the outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention includes 3 aspects (exercise, nutrition and breathing). Our intervention is a home-based multimodal prehabilitation program supported through an online platform.
  Interventions: Behavioral: Prehabilitation intervention
- Control (No Intervention): To support blinding, improve enrollment and reflect usual care, widely available physical activity (World Health Organization Recommendations for Physical Activity for ages 18-64 and >65) and healthy eating recommendations (Canada's Food Guide Snapshot) documents will be provided to control participants (without active or online support).

INTERVENTIONS:
Behavioral: Prehabilitation intervention — The intervention consists of exercise, nutritional support and breathing techniques. The exercise component consists of 1) strength training; 2) cardio and 3) stretching. Participants will be encouraged to complete self-directed and/or group sessions >= 3 times per week. Each intervention participant will be provided a unique login to the virtual prehabilitation platform, which is the STRIVE Trial website. The nutrition component includes: 1) protein supplementation; 2) nutrition advice to support healthy eating. For the breathing component, participants will be encouraged to watch the video on Inspiratory Muscle Training (IMT) which involves diaphragmatic breathing and coughing/huffing. They will also be provided with an instruction booklet to take to hospital with them to support postoperative conduct of IMT during early recovery.
  Arms: Intervention

SUMMARY:
The STRIVE Before Surgery Trial evaluates three pragmatic elements (recruitment, adherence, and follow-up) associated with participating in a home-based multimodal prehabilitation program supported through an online platform. Half of the participants will be randomized into the prehabilitation group, while the other half will be randomized into the control group.

DETAILED DESCRIPTION:
Background: The number of people presenting for surgery, and their risk profile, are increasing. People presenting for surgery face substantial risk of postoperative adverse events. Fifteen to 30% of patients suffer a serious medical or surgical complication after surgery, and 1 in 5 develop a new patient-reported disability that reflects a loss of independence in day-to-day life. More than 1.4 million inpatient surgical procedures are performed in Canada each year. Globally, >300 million surgical procedures occur annually. As an increasing number of people present for surgery, the average risk profile of this population is rising. Surgical patients are typically older and live with comorbidity. This means that strategies to improve patient outcomes and reduce resource utilization are urgently needed. Patients, the public, clinicians, and policy makers participating in 2 separate James Lind Alliance Priority Setting Partnerships (Canada & UK) identified prehabilitation as a Top 10 priority for perioperative research. Furthermore, prehabilitation is currently discussed in the popular media as a strategy to improve outcomes for the growing number of high-risk patients presenting for surgery.

Overarching Aim: The STRIVE Before Surgery Trial will evaluate three pragmatic elements (recruitment, adherence, and follow-up) that our experience in prehabilitation research demonstrate are necessary to support successful, large-scale evaluation. The investigators will concurrently use implementation science methodology to further refine processes for the larger trial. As this is a vanguard pilot trial, data from this trial will be combined with the future, large-scale trial.

Methods:

Design, setting and participants: The STRIVE Before Surgery Trial is an assessor blinded multicenter individual patient parallel-arm vanguard pragmatic randomized controlled trial.

People => 18 years old having inpatient abdominal, thoracic, pelvic, head-and-neck or vascular surgery with expected length of stay of => 2 days will be included.

Intervention: The intervention includes 3 aspects (exercise, nutrition and breathing). Our intervention is a home-based multimodal prehabilitation program supported through an online platform.

Outcomes and sample size: Primary outcomes are monthly recruitment, intervention adherence, retention, and elicitation of patient, clinician and researcher-identified barriers. Secondary outcomes are days at home in the 30 days after surgery, survival, length of stay, patient safety indicators, intensive care unit admission, non-home discharge, readmission, emergency department visits, and health system costs. Our vanguard trial sample size estimate is informed by a power calculation for the future large-scale trial. For the vanguard trial, a sample size of 144 directly links to our 3 feasibility outcomes: 1) recruitment of 144 participants over 8-10 months at our 5 sites will demonstrate our ability to average 2-4 participants per site per month. To continue the momentum of the trial, the pilot sample size can increase up to a maximum of 190 participants, providing time for the research team to seamlessly launch the full-scale trial. The pilot phase will merge into the full-scale trial. Having flexibility in the pilot sample size will support this process.

Expertise: Our team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected outcomes: Knowledge gained from our vanguard trial will directly inform the larger pragmatic trial, which will be powered to detect a minimally important difference in a patient-reported outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Scheduled, or on the pathway, for inpatient abdominal, thoracic, pelvic, head-and-neck or vascular surgery
3. Expected surgery date between 3 and 12 weeks from enrollment
4. Valid provincial health insurance number
5. Access to internet-enabled device
6. Email address

Exclusion Criteria:

1. Inability to read and communicate in English
2. Cognitive impairment preventing ability to provide informed consent independently
3. No telephone/cell phone
4. Cardiac, neurological or orthopedic procedure
5. Surgery with no curative intent (palliative surgery)
6. Patient not interested in participating in the context of their Telephone Assessment of Physical Activity (TAPA) score
7. Any of the following cardiovascular conditions:

   1. Severe valvular heart disease that limits a patient's ability to ambulate on level ground, or is associated with syncope or dyspnea
   2. Severe cardiac dysrhythmias that limit a patient's ability to ambulate on level ground, or is associated with syncope or dyspnea
   3. Recent myocardial infarction (within 6 weeks prior to enrollment - based on the Heart and Stroke Foundation's Heart Walk program)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Monthly recruitment | 1 year
  Recruited patients per center per month will be analyzed descriptively to generate a mean and standard deviation. Recruitment feasibility will be judged based on criteria pre-established that consider the number of available, committed sites in Ontario.
Intervention adherence | pre-surgery
  The proportion of prescribed prehabilitation tasks adhered to
Retention | 1 month, year 1
  The proportion of participants retained at 30-day patient-reported follow up will be calculated with a 95% confidence interval based on Wilson's method.
Elicitation of patient, clinician and researcher-identified barriers | 1 year
  For each target group, the frequency of domains identified as barriers will be calculated.
Patient-reported disability using the World Health Organization Disability Assessment Schedule 2.0 (WHODAS) (to be merged with larger trial) | 1 month, 3 month, 1 year
  The WHODAS is a patient-reported disability scale that assesses limitations in six major life domains (i.e., cognition, mobility, self-care, social interaction, life activities, participation in society). Each questionnaire item is scored on a Likert scale ranging from 0 to 4. The sum of the responses is the WHODAS Disability Score (range: 0 to 48), which is expressed as a percentage of the maximum possible score

SECONDARY OUTCOMES:
Days at home (to be merged with larger trial) | 1 month, 1 year
  A count of days at home in the 30-days after surgery is a validated patient-centered outcome that can be ascertained from routinely collected data
Survival (to be merged with larger trial) | 1 year
  All cause deaths and survival time in the 30-days and year after surgery will be captured from vital statistics
Length of Stay (to be merged with larger trial) | 1 year
  Days from surgical admission to discharge
Patient Safety Events (to be merged with larger trial) | 1 year
  A validated set of in-hospital patient safety indicators will be captured from the index hospitalization record
Intensive care unit admission (to be merged with larger trial) | 1 year
  Intensive care unit admission captured by administrative data
Non-home discharge (to be merged with larger trial) | 1 year
  Discharge from the index hospitalization via transfer to a non-home location or death
Re-admission (to be merged with larger trial) | 1 month, 1 year
  Number of re-admissions to hospital
Emergency department visits (to be merged with larger trial) | 1 month, 1 year
  Number of emergency department visits
Health system costs (to be merged with larger trial) | 1 month, 1 year
  A validated patient-level costing algorithm will be used to capture all health system costs accrued within 30-days and 1-year after surgery
Health Related Quality of Life using the EQ-5D-5L (to be merged with larger trial) | 1 month, 3 month, 1 year
  EQ-5D-5L will be used to capture health related quality of life at baseline, pre-op, 30, 90, and 365 days after surgery.
In-hospital complications | Up to 1 month
  Postoperative Morbidity Survey (POMS) is a tool used to used to identify complications. At time of discharge, participants will be administered a patient-reported version of the POMS tool

CONTACTS AND LOCATIONS:
Overall Officials: Daniel McIsaac, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.

REFERENCES:
- [Derived] McIsaac DI, Tandon P, Kidd G, Branje K, Hladkowicz E, Hallet J, Wijeysundera DN, Lee S, McNeely ML, Taljaard M, Gillis C; STRIVE Trial Investigators; Canadian Perioperative Anesthesia Clinical Trials Group (PACT). STRIVE pilot trial: a protocol for a multicentre pragmatic internal pilot randomised controlled trial of Structured TRaining to Improve fitness in a Virtual Environment (STRIVE) before surgery. BMJ Open. 2024 Nov 7;14(11):e093710. doi: 10.1136/bmjopen-2024-093710. PMID 39510784